CLINICAL TRIAL: NCT01086358
Title: A Single Center Randomized Open-Label Two Arm Crossover Study of Subject Productivity Improvement and Satisfaction With Migraine Treatment Using Treximet vs Usual Triptan
Brief Title: Does Treximet Improve Productivity and Patient Satisfaction Due to Sustained Response and Consistency of Response?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: GlaxoSmithKline (Industry); Currax Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jennifer Kriegler, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 09-602
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Workplace Migraine Treatment
Keywords: Productivity; Migraine; Treximet; Triptan
MeSH Terms: conditions — Migraine Disorders | interventions — Tryptamines; Sumatriptan; sumatriptan-naproxen; Naproxen

STUDY DESIGN:
Intervention Model Description: This was a randomized, open-label, 6-attack (3-attacks per arm) crossover design in which subjects were randomized to threat their first 3 workplace migraines with sumatriptan/naproxen sodium or with their usual triptan monotherapy before treating their subsequent 3 workplace migraines with the opposite medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Triptan (Active Comparator): Arm 1 subjects began with their prescribed triptan
  Interventions: Drug: Triptan
- Treximet 85Mg-500Mg Tablet (Active Comparator): Arm 2 subjects began with Treximet (sumatriptan 85 mg/naproxen sodium 500 mg)
  Interventions: Drug: Treximet 85Mg-500Mg Tablet

INTERVENTIONS:
Drug: Triptan — Usual prescribed triptans may include:sumatriptan, rizatriptan, naratriptan, almotriptan, eletriptan, zolmitriptan
  Other Names: Sumatriptan,rizatriptan,naratriptan,almotriptan,eletriptan,zolmitriptan
  Arms: Triptan
Drug: Treximet 85Mg-500Mg Tablet — Treximet is 85 mg sumatriptan plus 500 mg naproxen sodium
  Other Names: Sumatriptan 85 mg plus naproxen sodium 500 mg
  Arms: Treximet 85Mg-500Mg Tablet

SUMMARY:
Researchers want to learn about work productivity after treatment of a migraine headache with your usual migraine medication as compared to your work productivity after treatment with Treximet.

During this research subjects will take Treximet to treat 3 workday migraine attacks. For a second part of the research subjects will take their usual prescribed medication for 3 workday migraine attacks. The subjects will complete questionnaires after treating each migraine.

DETAILED DESCRIPTION:
A subject who is identified for study participation will participate in the screening and enrollment visit which determines the migraine treatment arm to which the subject will be randomized first. The subject will have a physical exam, vital signs recorded, health and medication questions asked, questionnaires completed and a headache diary explained and dispensed to the subject. If the subject is randomized to the Treximet treatment arm during the first part of the study, Treximet will be dispensed for use in treating workday migraines.

The subject will call the study coordinator after treating a workday migraine and will report information about the migraine to the coordinator. When the subject has treated and reported on 3 migraines, the interim visit will be scheduled. The subject will bring the study diary and Treximet containers (if this was the arm the subject completed)to this visit. The subject will be asked about adverse events and medication changes as well as confirmation and review of the completed questionnaires and diaries from the prior weeks of study participation. The subject will be given new diaries and questionnaires (and Treximet to use if usual prescribed triptan was the treatment in the first arm) and repeat the activities to treat 3 more workday migraines.

When the subject has notified the study coordinator about treating the 3rd workday migraine in this part of the study, the subject will be scheduled for the final study visit. The subject will bring the completed migraine diaries, completed questionnaires (and Treximet bottles if used during this arm) to the study visit. The subject will have the diaries and questionnaires reviewed, be asked about adverse events and medication changes and complete the final study questionnaires at this visit.

ELIGIBILITY:
Inclusion Criteria:

* episodic migraine diagnosis
* age 18 or older
* currently using a triptan as primary migraine monotherapy
* currently employed
* if of childbearing potential, willing to prevent pregnancy during study participation
* able to understand and consent to study participation

Exclusion Criteria:

* younger than age 18
* not having episodic migraine diagnosis
* not using a triptan as primary migraine monotherapy
* not currently employed
* pregnant or nursing or unwilling to prevent pregnancy during study participation
* unable to understand and consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Kriegler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, 9500 Euclid Avenue, C-21, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Mathew NT, Landy S, Stark S, Tietjen GE, Derosier FJ, White J, Lener SE, Bukenya D. Fixed-dose sumatriptan and naproxen in poor responders to triptans with a short half-life. Headache. 2009 Jul;49(7):971-82. doi: 10.1111/j.1526-4610.2009.01458.x. Epub 2009 May 27. PMID 19486178
- [Background] Dowson AJ, Tepper SJ, Baos V, Baudet F, D'Amico D, Kilminster S. Identifying patients who require a change in their current acute migraine treatment: the Migraine Assessment of Current Therapy (Migraine-ACT) questionnaire. Curr Med Res Opin. 2004 Jul;20(7):1125-35. doi: 10.1185/030079904125004079. PMID 15265257
- [Background] Cleves C, Tepper SJ. Sumatriptan/naproxen sodium combination for the treatment of migraine. Expert Rev Neurother. 2008 Sep;8(9):1289-97. doi: 10.1586/14737175.8.9.1289. PMID 18759540
- [Background] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 Subjects who are employed in a paying job, who have episodic migraine (<15 days/month), who are using an acute care triptan monotherapy for their migraine (excluding combinations of any sort, such as acetaminophen [APAP] and non-steoridals [NSAIDs]) and who have no contraindications to triptan or NSAID use.
Pre-assignment Details: This study had no wash-out or run-in phase.
Groups:
- Usual Prescribed Triptan First: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule. To account for the correlation from patients acting as their own controls in this crossover design, a standard deviation of the difference equal to 2.5 is assumed. Under these assumptions, a total sample of 60, with 30 in each sequence, would power the study at 86%.
- Treximet Arm First: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule.
  Treximet for migraine treatment: Treximet is the combination of sumatriptan 85 mg plus naproxen sodium 500mg. To account for the correlation from patients acting as their own controls in this crossover design, a standard deviation of the difference equal to 2.5 is assumed. Under these assumptions, a total sample of 760, with 30 in each sequence, would power the study at 86%.
Period: First Intervention
Arm/Group | Usual Prescribed Triptan First | Treximet Arm First
Started | 30 (30 subjects enrolled.) | 29 (30 subjects enrolled, 1 withdrew before randomization)
Completed | 21 | 24
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 9 | 4
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Usual Prescribed Triptan First | Treximet Arm First
Started | 21 | 24
Completed | 17 | 20
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- All Completed Study Participants: Participants received their usual prescribed triptan or Treximet, depending on the randomization schedule.
  Usual prescribed triptan: usual prescribed triptans may include:sumatriptan, rizatriptan, naratriptan, almotriptan, eletriptan, zolmitriptan
Arm/Group | All Completed Study Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects were lost to follow-up or withdrew consent.
  years | 41.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all subjects completed both study arms.
  Participants
    Female | 33
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 37 patients completed both phases of the study and make up the primary data set.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 34
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Workplace Productivity and Activity Impairment Scale (WPAI).
Description: The primary outcome measure was lost productivity (workplace productivity + non-workplace activity time) as measured by a variant of the Work Productivity and Activity Impairment Scale (WPAI) at 6 months. The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The unit of analysis is hours lost. The higher the score the greater impact on productivity. The range depends on the length of the attack, but in the sample among all observed attacks, lost work productivity ranged from 0-10.5 hours, while lost non-workplace activity time ranged from 0 to 8.95 hours. The total lost productivity is the sum of lost work productivity and lost non-workplace activity time.
Time Frame: 6 months
Population: This includes all patients that completed all study visits are included in this efficacy analysis
Measure: Mean (95% Confidence Interval); unit: hours
Groups:
- Arm 1 - Triptan: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule.
  Arm 1 Triptan: Usual prescribed triptans may include:sumatriptan, rizatriptan, naratriptan, almotriptan, eletriptan, zolmitriptan
- Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule.
  Arm 2 - Sumatriptan/naproxen sodium (Treximet): Treximet is the combination of sumatriptan 85 mg plus naproxen sodium 500mg
Arm/Group | Arm 1 - Triptan | Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm
Number analyzed (Participants) | 37 | 37
hours | 4.15 [2.93 to 5.36] | 2.44 [1.23 to 3.65]
Statistical Analysis 1: Comparison: Arm 1 - Triptan vs Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm; Analysis is a superiority comparison based on the use of linear mixed effect model with subject as a random effect, with treatment as the primary fixed effect and including study period and treatment order as other fixed effects; Test type: Superiority; p = 0.007, Mixed Models Analysis; As noted above, results are adjusted for study period and treatment order; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.92 to -0.49]

2. Secondary Outcome: Lost Workplace Productivity
Description: This outcome measure was lost workplace productivity as measured by a variant of the Work Productivity and Activity Impairment Scale (WPAI) at 6 months.The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The unit of analysis is hours lost. The higher the score the greater impact on productivity. The range depends on the length of the attack, but in the sample among all observed attacks, lost work productivity ranged from 0-10.5 hours, while lost non-workplace activity time ranged from 0 to 8.95 hours. The total lost productivity is the sum of lost work productivity and lost non-workplace activity time.
Time Frame: 6 months
Population: This includes all patients that completed all study visits are included in this efficacy analysis
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1 - Triptan | Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm
Number analyzed (Participants) | 37 | 37
hours | 2.25 [1.60 to 2.90] | 1.23 [0.58 to 1.87]
Statistical Analysis 1: Comparison: Arm 1 - Triptan vs Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.010, Mixed Models Analysis; As noted above, results are adjusted for study period and treatment order; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.79 to -0.27]

3. Secondary Outcome: Lost Activity Time
Description: This outcome measure was lost activity time as measured by a variant of the Work Productivity and Activity Impairment Scale (WPAI) at 6 months.The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The unit of analysis is hours lost. The higher the score the greater impact on productivity. The range depends on the length of the attack, but in the sample among all observed attacks, lost work productivity ranged from 0-10.5 hours, while lost non-workplace activity time ranged from 0 to 8.95 hours. The total lost productivity is the sum of lost work productivity and lost non-workplace activity time.
Time Frame: 6 Months
Population: This includes all patients that completed all study visits are included in this efficacy analysis
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1 - Triptan | Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm
Number analyzed (Participants) | 37 | 37
hours | 1.89 [1.19 to 2.60] | 1.22 [0.51 to 1.92]
Statistical Analysis 1: Comparison: Arm 1 - Triptan vs Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.059, Mixed Models Analysis; As noted above, results are adjusted for study period and treatment order; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.39 to 0.03]

4. Secondary Outcome: Favorable Response on Migraine-ACT
Description: The Migraine-ACT is a 4-item scale with yes/no responses. A score of 3 or more is considered favorable. The primary efficacy dataset included the 37 patients that completed both phases of the study and uses the last observed headache. The Migraine-ACT is reported as a binary measure (3 or more positive responses). The outcome presented included the percentage with a score of 3 or more, and the Odds ratio comparing the two treatments.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of favorable responses
Arm/Group | Arm 1 - Triptan | Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm
Number analyzed (Participants) | 37 | 37
percentage of favorable responses | 46 [30 to 63] | 71 [54 to 84]
Statistical Analysis 1: Comparison: Arm 1 - Triptan vs Arm 2 - Sumatriptan/Naproxen Sodium (Treximet) Arm; Logistic regression models with generalized estimating equations were used. In these models, a logit link function was used for a favorable response (yes/no) with treatment as the primary fixed effect and including study period and treatment order as other fixed effects; Test type: Superiority; p = 0.016, Regression, Logistic; As noted above, results are adjusted for study period and treatment order; Odds Ratio (OR) = 2.89, 95% CI 2-sided [1.22 to 6.84]

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Description: Adverse events were noted from the date of the first study visit until the end of study visit was completed, grouped by the treatment medication in use. There were no serious AEs. 45 patients entered the Triptan arm and 45 patients entered the Treximet arm. 12 patients failed to report AE status and were considered to be free from AEs in the calculations below.
Groups:
- Usual Prescribed Triptan: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule. To account for the correlation from patients acting as their own controls in this crossover design, a standard deviation of the difference equal to 2.5 is assumed. Under these assumptions, a total sample of 760, with 30 in each sequence, would power the study at 86%.
- Treximet Arm: Subjects will be randomized to either of two arms at enrollment in this study. They may start with their usual prescribed triptan or Treximet, depending on the randomization schedule.
  Treximet for migraine treatment: Treximet is the combination of sumatriptan 85 mg plus naproxen sodium 500mg. To account for the correlation from patients acting as their own controls in this crossover design, a standard deviation of the difference equal to 2.5 is assumed. Under these assumptions, a total sample of 760, with 30 in each sequence, would power the study at 86%.
Arm/Group | Usual Prescribed Triptan | Treximet Arm
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 18/45 | 15/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Prescribed Triptan (N=45) | Treximet Arm (N=45)
Somnolence (Nervous system disorders) | 8 | 4 — Sleepiness
Nausea (Gastrointestinal disorders) | 5 | 6
Lightheadedness (Nervous system disorders) | 4 | 1 — Lightheaded, head pressure and tightness and head rush, diaphoresis
Fatigue (General disorders) | 4 | 1
Chest Discomfort (General disorders) | 1 | 1
Giddiness (Nervous system disorders) | 1 | 1 — Loopiness and Dopey
Apraxia (Nervous system disorders) | 1 | 1 — Word finding difficulty
Bladder pain (Renal and urinary disorders) | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Xerostomia (General disorders) | 2 | 0 — dry mouth and jaw tightness
Paresthesia (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Unusually high number of subjects lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT01086358/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT01086358/ICF_001.pdf